CLINICAL TRIAL: NCT01409668
Title: Efficacy of Two Yogurt Formulations as Health Promoting Agents in Healthy Humans
Brief Title: Efficacy of Two Yogurt Formulations in Healthy Humans
Acronym: MPH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Micropharma Limited (Industry)
Responsible Party: Dr. Peter Jones, Director of RCFFN, RCFFN, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2007:070
Record Dates: First submitted 2011-06-22; First posted 2011-08-04 (Estimated); Last update posted 2011-08-04 (Estimated); Status verified 2007-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L. Amylovorus (Experimental)
  Interventions: Dietary Supplement: L. Amylovorus
- L. Fermentum (Experimental)
  Interventions: Dietary Supplement: L. Fermentum

INTERVENTIONS:
Dietary Supplement: L. Amylovorus — L. Amylovorus
  Arms: L. Amylovorus
Dietary Supplement: L. Fermentum — L. Fermentum
  Arms: L. Fermentum

SUMMARY:
This study is to evaluate the safety and efficacy of consumption of: L.Ruteri containing yogurt, L.Fermentum containing yogurt VERSUS placebo on plasma lipids, as well as gastrointestinal microflora distribution in hyperlipidemic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* aged 18-60 yr
* plasma LDL-C 130-260 mg/dl
* TG levels below 400 mg/dl
* body mass index (BMI) rangewill be 22 to 32 kg/m2
* permitted to take stable doses of thyroid hormone and anti hypertensive agents, as long as these are continued equivalently throughout the duration of study

Exclusion Criteria:

* history of recent (i.e. less than 3 mo) or chronic use of oral hypolipidemic therapy, including fish oils, or probucol within the last 6 mo, - history of chronic use of alcohol (>2 drinks/d), systemic antibodies, corticosteroids, androgens, or phenytoin,
* myocardial infarction, coronary artery bypass, or other major surgical procedures within the last six months
* recent onset of angina, congestive heart failure, inflammatory bowel disease, pancreatitis, diabetes, lactose intolerance or significant current (ie. onset within past three months) gastrointestinal, renal, pulmonary, hepatic or biliary disease, or cancer (evidence of active lesions, chemotherapy or surgery in the past year
* chronic user of probiotics, fiber laxative (greater than 2 doses/wk), or stimulant laxatives or has a history of eating disorders, exercise greater than 15 miles/wk or 4,000 kcal/wk.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Cholesterol Metabolism | 1 month